CLINICAL TRIAL: NCT02178670
Title: Study of Cancer Stem Cell Vaccine That as a Specific Antigen in Metastatic Adenocarcinoma of the Ovarian
Brief Title: Safety and Effectivity Immunotherapy to Treat Ovarian Cancer With Cancer Stem Cells Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLO-001; 201401 (Other Grant/Funding Number: The research fund of Fuda cancer hospital in Guangzhou)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2014-06

CONDITIONS: Neoplasms,Ovarian
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-cancer stem cell vaccine (Placebo Comparator): There is no cancer stem cell vaccine in this group
  Interventions: Biological: CSC-DC
- giving low dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: CSC-DC
- giving middle dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: CSC-DC
- giving high dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: CSC-DC

INTERVENTIONS:
Biological: CSC-DC

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinct murine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring antitumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with ovarian Cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the ovarian cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the ovarian cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-ovarian cancer CSC immunity induced by ovarian cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of ovarian cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with ovarian cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

Patients with epithelial ovarian cancer FIGO (Fédération Internationale de Gynécologie et d'Obstétrique) stage III in remission after treatment with surgery (hysterectomy and ovariectomy) and after the first primary chemotherapy (standard treatment e.g. 6-9x Carboplatin/Taxane)

1. Age > 18 ≤ 75 years
2. Histological confirmed FIGO stage III ovarian epithelial cancer
3. Stable disease at screening visit: negative CT and CA-125 within normal range
4. Karnofsky status ≥ 70% and/or ECOG (Eastern Cooperative Oncology Group) performance status 0-2
5. Life expectancy ≥ 6 months
6. Adequate hematological function (WBC (white blood cells) ≥ 3000/µl, hemoglobin ≥ 10.0 g/dL, platelets > 100,000/µl)
7. Adequate renal and hepatic function (serum creatinine ≤ 2.0 mg/dL, bilirubin total < 2 mg/dL, PT (INR) ≤ 1.5x institutional upper limit of normal)
8. Signed and dated informed consent before the start of any study-specific procedure
9. Body weight > 50 kg

Exclusion Criteria:

1. Surgery, radiation therapy or chemotherapy within eight weeks prior to leukapheresis
2. Other biological therapy (Interferons, TNF (Tumor necrosis factors), Interleukins, mABs (Monoclonal antibodies), biological response modifiers) within eight weeks prior to undergo the leukapheresis
3. History or presence of systemic autoimmune disease (such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma or multiple sclerosis)
4. Participation in other clinical trials or treatments with an investigational drug within four weeks prior to enrollment
5. Serious intercurrent chronic or acute illness such as severe asthma or COPD (Chronic Obstructive Pulmonary Disease), cardiac (NYHA (New York Heart Association ) class III or IV) or hepatic disease, or other illness considered to constitute an unwarranted high risk for investigational drug treatment
6. History of another malignancy within five years prior to study enrollment, except curatively treated non-melanotic skin cancer or cervical cancer in situ
7. Presence of an active acute or chronic infection, including syphilis, HIV or viral hepatitis B and/or C
8. Current treatment with corticosteroids (except of local) or other immunosuppressive agents such as azathioprine or cyclosporine A is excluded on the basis of its potential immune suppression. Any systemic steroid therapy must have been discontinued six weeks prior to undergo the leukapheresis
9. Patients who have undergone organ transplantation
10. Legally incapacitated persons and/or other circumstances, which make it difficult for the subject to understand the nature, meaning and consequences of the clinical study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary study purpose to determine the safety of immunization with cancer stem cells vaccine by the number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccine immune responses to the immunizations by the data of body measurements | 1 month
  The secondary objectives are to evaluate the vaccine immune responses including cellular immunity and humoral immunity

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/